CLINICAL TRIAL: NCT01350999
Title: A Phase 3 Long-term Study of TAK-085 in Subjects With Hypertriglyceridemia
Brief Title: Long-term Efficacy and Safety Study of TAK-085 in Participants With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-085/OCT-001; JapicCTI-090936 (Registry Identifier: JapicCTI); U1111-1120-7892 (Registry Identifier: WHO); JapicCTI-R140451 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Hypertriglyceridemia
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertriglyceridemia | interventions — TAK-085; Omacor; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-085 2 g (Experimental): TAK-085 2 g, orally, once daily for up to 52 weeks.
  Interventions: Drug: omega-3-acid ethyl esters 90 (TAK-085)
- TAK-085 4 g (Experimental): TAK-085 2 g, orally, twice daily for up to 52 weeks.
  Interventions: Drug: omega-3-acid ethyl esters 90 (TAK-085)
- EPA-E 1.8 g (Active Comparator): Eicosapentaenoic acid-ethyl (EPA-E) capsule 0.6 g, orally, three-times daily for up to 52 weeks.
  Interventions: Drug: Eicosapentaenoic acid-ethyl (EPA)

INTERVENTIONS:
Drug: omega-3-acid ethyl esters 90 (TAK-085) — Omega-3-acid ethyl esters 90 (TAK-085) capsules. Each one gram of fatty acid in TAK-085 contains approximately 465 mg of EPA plus 375 mg of docosahexaenoic acid-ethyl as ethyl esters.
  Other Names: LOVAZA; Omacor
  Arms: TAK-085 2 g; TAK-085 4 g
Drug: Eicosapentaenoic acid-ethyl (EPA) — EPA-E capsules
  Arms: EPA-E 1.8 g

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TAK-085, once daily (QD) or twice daily (BID), compared to ethyl eicosapentaenoate (EPA-E), three times daily (TID) in participants with hypertriglyceridemia undergoing lifestyle modification.

DETAILED DESCRIPTION:
TAK-085 is an oral capsule medicine licensed to Takeda Pharmaceutical Company Ltd. TAK-085 contains omega-3 fatty acid ethyl (mainly, ethyl eicosapentaenoate (EPA-E) and ethyl docosahexaenoic acid (DHA-E)).

This is a phase 3, open-label, randomized study to evaluate the efficacy and safety of TAK-085. In addition, EPA-E is also administered for 52 weeks for reference to evaluate the safety of TAK-085 in participants with hypertriglyceridemia who are undergoing lifestyle modification.

The study period is a total of 56 weeks, comprised of a 4- week screening period and 52 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Visit 1 (Week -4)

1. Undergoing lifestyle modification.
2. Triglyceride (TG) level (fasting state) 150 mg/dL or higher and less than 750 mg/dL at Visit 1 (Week -4).
3. Both genders, aged from 20 to less than 75 years at the time of signing informed consent.
4. Outpatient.
5. Capable of understanding and complying with protocol requirements.
6. Signed a written, informed consent form prior to the initiation of any study procedures.
7. A female with childbearing potential (premenopausal and non-sterilized) must have agreed to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

   Visit 2 (Week -2)
8. Fasting TG level 150 mg/dL or higher and less than 750 mg/dL at Visit 2 (Week -2).
9. Difference in fasting low density lipoprotein-cholesterol (LDL-C) level between Visit 1 (Week -4) and Visit 2 (Week -2) within 25% of the higher value

Exclusion Criteria:

Visit 1 (Week -4)

1. Any coronary artery diseases (CAD, e.g., confirmed myocardial infarction and angina pectoris) within 6 months prior to Visit 1 (Week -4) or a history of revascularization.
2. Received aortic aneurysmectomy or had had aortic aneurysm within 6 months prior to Visit 1 (Week -4).
3. History or complication of a clinically significant hemorrhagic disease (e.g., hemophilia, capillary fragility illness, digestive tract ulcer, urinary tract haemorrhage, hemoptysis, vitreous haemorrhage) within 6 months prior to Visit 1 (Week -4).
4. Diagnosed with pancreatitis.
5. Diagnosed with lipoprotein lipase (LPL) deficiency, apolipoprotein C-II deficiency or type III familial hyperlipidemia.
6. Cushing's syndrome, uremia, systemic lupus erythematosus (SLE) or serum dysproteinemia.
7. Type 1 diabetes mellitus or with uncontrolled type 2 diabetes mellitus defined by glycosylated hemoglobin (HbA1C) level of 8.0% or higher at Visit 1 (Week -4).
8. Stage III hypertension defined by systolic blood pressure of 180 mmHg or higher or diastolic blood pressure of 110 mmHg or higher regardless of the use of antihypertensive medication.
9. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level at Visit 1 (Week -4) was not less than twice the upper limit of the normal reference range.
10. If female, was pregnant or lactating.
11. Habitual drinking defined by an average daily alcohol intake of 100 mL or more , drug abuse or drug dependency, or a history of any of these conditions.
12. Started to take any antihyperlipidemic drugs within 4 weeks prior to Visit 1 (Week -4).
13. Received any investigational products (including those for post-marketing clinical study) within 12 weeks prior to Visit 1 (Week -4).
14. Received TAK-085 in a clinical study.
15. Judged as being ineligible for study participation by the investigator or subinvestigator for any other reasons.

    Visit 2 (Week -2)
16. ALT or AST level at Visit 2 (Week -2) was twice the upper limit of the normal reference range or higher.
17. Needed a change in the dose of antihyperlipidemic drugs or antidiabetic drugs, addition of a new drug or a change in the type of the drugs during the screening period.
18. Judged as being ineligible for study participation by the investigator or subinvestigator for any other reasons.

    Visit 3 (Week 0)
19. Needed a change in the dose of antihyperlipidemic drugs or antidiabetic drugs, addition of a new drug or a change in the type of the drugs during the screening period.
20. Judged as being ineligible for study participation by the investigator or subinvestigator for any other reasons

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor, Clinical Cell Biology and Medicine, Study Director — Graduate School of Medicine, Chiba University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 50 investigative sites in Japan from 11 November 2009 to 11 January 2011.
Pre-assignment Details: Participants with hypertriglyceridemia were randomized to receive omega-3-acid ethyl esters 90 (TAK-085) 2 g once daily or TAK-085 2 g twice daily or EPA-E 0.6 g three-times daily.
Groups:
- TAK-085 2 g: TAK-085 2 g capsule, orally, once daily for up to 52 weeks.
- TAK-085 4 g: TAK-085 2 g capsules, orally, twice daily for up to 52 weeks.
Period: Overall Study
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Started | 165 | 171 | 167
Treated | 165 | 171 | 167
Completed | 157 | 157 | 146
Not Completed | 8 | 14 | 21
Not completed — Adverse Event | 4 | 9 | 10
Not completed — Voluntary withdrawal | 3 | 4 | 6
Not completed — Difficulty Making it to Study Visit | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g | Total
Number analyzed (Participants) | 165 | 171 | 167 | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.95) | 55.9 (10.12) | 55.8 (9.27) | 55.9 (10.11)
Age, Customized [Number; unit: participants]
  ≥20 - <65 years | 119 | 134 | 136 | 389
  ≥65 - ≤74 years | 46 | 37 | 31 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 48 | 145
  Male | 118 | 121 | 119 | 358
Region of Enrollment [Number; unit: participants]
  Japan | 165 | 171 | 167 | 503
Menopause Status [Number; unit: participants]
  Yes | 38 | 42 | 39 | 119
  No | 5 | 7 | 5 | 17
  Unknown | 4 | 1 | 4 | 9
  Not Applicable | 118 | 121 | 119 | 358
Height, Categorical [Number; unit: participants]
  <160 cm | 48 | 45 | 48 | 141
  ≥160 - <170 cm | 67 | 77 | 66 | 210
  ≥170 cm | 50 | 49 | 53 | 152
Height [Mean (Standard Deviation); unit: cm] | 164.2 (9.40) | 164.0 (8.69) | 164.4 (9.65) | 164.2 (9.23)
Weight, Categorical [Number; unit: participants]
  <60 kg | 32 | 34 | 32 | 98
  ≥60.0 - <70.0 kg | 57 | 53 | 43 | 153
  ≥70.0 - <80.0 kg | 44 | 50 | 57 | 151
  ≥80.0 kg | 32 | 34 | 35 | 101
Weight [Mean (Standard Deviation); unit: kg] | 70.02 (12.291) | 70.46 (12.097) | 71.61 (13.311) | 70.70 (12.568)
Body Mass Index, Categorical [Number; unit: participants]
  <25.0 kg/m^2 | 77 | 72 | 60 | 209
  ≥25.0 - <30.0 kg/m^2 | 71 | 74 | 83 | 228
  ≥30.0 kg/m^2 | 17 | 25 | 24 | 66
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.90 (3.673) | 26.11 (3.526) | 26.33 (3.301) | 26.12 (3.500)
Smoking Classification [Number; unit: participants]
  Never Smoked | 59 | 56 | 47 | 162
  Current Smoker | 52 | 47 | 58 | 157
  Ex-Smoker | 54 | 68 | 62 | 184
Waist Circumference, Categorical [Number; unit: participants]
  Male <85.0 cm | 22 | 29 | 19 | 70
  Male ≥85.0 cm | 96 | 92 | 100 | 288
  Female <90.0 cm | 26 | 30 | 26 | 82
  Female ≥90.0 cm | 21 | 20 | 22 | 63
Waist Circumference [Mean (Standard Deviation); unit: cm] | 90.39 (8.607) | 90.75 (9.169) | 91.16 (9.284) | 90.77 (9.015)
Coronary Artery Disease (CAD) Category [Number; unit: participants] — CAD Patient Categories define the degree of risk of CAD according to Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases. Categories are classified by the degree of risks in the patient [e.g, smoking, hypertension, excluding level of low density lipoprotein cholesterol (LDL-C)]. Category I=Low risk (best), Category II=Middle risk, Category III=High Risk and History of CAD.
  participants
    Category I | 7 | 9 | 3 | 19
    Category II | 70 | 71 | 56 | 197
    Category III | 86 | 86 | 102 | 274
    History of CAD | 2 | 5 | 6 | 13
Hypertension [Number; unit: participants]
  Yes | 110 | 115 | 115 | 340
  No | 55 | 56 | 52 | 163
Diabetes Mellitus (Including Impaired Glucose Tolerance) [Number; unit: participants]
  Yes | 50 | 63 | 71 | 184
  No | 115 | 108 | 96 | 319
Low High Density Lipoprotein - Cholesterol (HDL-C) [Number; unit: participants]
  Yes | 42 | 39 | 45 | 126
  No | 123 | 132 | 122 | 377
Administration of 3-hydroxy 3-methylglutaryl coenzyme A (HMGCoA) Reductase Inhibitor [Number; unit: participants]
  Yes | 64 | 66 | 65 | 195
  No | 101 | 105 | 102 | 308
Triglycerides, Categorical [Number; unit: participants] — The number of participants with available triglyceride data are 164, 169 and 167 in each treatment arm, respectively.
  participants
    <150 mg/dL | 16 | 12 | 14 | 42
    ≥150 - <300 mg/dL | 103 | 107 | 109 | 319
    ≥300 - <500 mg/dL | 38 | 43 | 37 | 118
    ≥500 mg/dL | 7 | 7 | 7 | 21
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — The number of participants with available triglyceride data are 164, 169 and 167 in each treatment arm, respectively.
  mg/dL | 254.7 (97.80) | 270.0 (101.19) | 264.2 (111.62) | 263.0 (103.71)
Low Density Lipoprotein - Cholesterol (LDL-C), Categorical [Number; unit: participants]
  <140 mg/dL | 101 | 116 | 102 | 319
  ≥140 mg/dL | 64 | 55 | 65 | 184
Low Density Lipoprotein - Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 133.2 (29.85) | 129.0 (30.26) | 129.3 (33.00) | 130.5 (31.06)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: 52 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
participants | 106 | 110 | 109

2. Primary Outcome: Number of Participants With TEAEs Associated With Abnormal Changes in Vital Signs
Time Frame: 52 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
participants | 0 (12.58) | 0 (12.64) | 0 (12.80)

3. Primary Outcome: Number of Participants With TEAEs Associated With Abnormal Changes in Body Weight
Time Frame: 52 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
participants | 0 (0.907) | 0 (0.870) | 0 (0.919)

4. Primary Outcome: Number of Participants With Clinically Significant Findings in Electrocardiogram After Study Drug Administration
Description: Participants whose results of electrocardiograms were judged as abnormal and clinically significant by investigator after study drug administration were counted in this measure.
Time Frame: 52 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Categorized Into Investigations System Organ Class (SOC) Related to Chemistry, Hematology or Urinalysis
Time Frame: 52 Weeks
Population: Safety Analysis Set included all participants who received at least one dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
participants | 24 | 21 | 23

6. Secondary Outcome: Percent Change From Baseline in Triglyceride Level
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set (all participants who were randomized and received at least one dose of the investigational product) with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
percent change
  Week 4 (n=163, 168, 166) | -10.875 (28.1914) | -24.550 (26.7987) | -5.743 (35.8469)
  Week 8 (n=162, 166, 163) | -10.474 (36.1225) | -26.555 (24.1354) | -5.796 (36.2369)
  Week 12 (n=162, 166, 161) | -11.628 (28.6330) | -21.689 (27.9188) | -9.204 (34.5555)
  Week 16 (n=160, 165, 161) | -9.363 (35.5523) | -20.735 (35.0625) | -9.522 (36.2768)
  Week 20 (n=161, 164, 157) | -12.965 (29.2649) | -21.483 (28.1817) | -7.400 (37.9737)
  Week 24 (n=158, 162, 155) | -13.393 (34.8938) | -23.863 (31.2129) | -8.269 (38.8420)
  Week 28 (n=159, 159, 153) | -12.644 (33.3250) | -25.119 (31.4602) | -9.422 (34.4423)
  Week 32 (n=159, 160, 151) | -11.464 (36.7968) | -27.219 (27.8708) | -9.867 (36.9807)
  Week 36 (n=156, 158, 151) | -16.190 (33.2777) | -26.535 (27.0283) | -9.616 (42.1895)
  Week 40 (n=159, 158, 151) | -13.934 (35.8353) | -25.062 (30.7020) | -15.345 (33.6494)
  Week 44 (n=158, 156, 149) | -17.156 (31.8849) | -24.402 (30.1719) | -12.363 (38.4921)
  Week 48 (n=156, 155, 147) | -14.722 (33.1045) | -26.478 (31.4535) | -10.185 (39.0040)
  Week 52 (n=153, 151, 145) | -14.219 (31.1401) | -26.023 (28.3644) | -13.872 (40.9936)

7. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein - Cholesterol (LDL-C)
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
percent change
  Week 4 (n=165, 170, 167) | -2.219 (14.5984) | -2.327 (17.3965) | -3.018 (16.3629)
  Week 8 (n=164, 168, 165) | -2.890 (15.7779) | -3.209 (17.1870) | -4.423 (16.7481)
  Week 12 (n=163, 168, 161) | -4.692 (15.5025) | -4.778 (16.2444) | -4.542 (16.6098)
  Week 16 (n=163, 167, 161) | -4.689 (17.3729) | -4.404 (18.8456) | -4.551 (17.6688)
  Week 20 (n=162, 166, 157) | -4.953 (16.1426) | -3.088 (17.7755) | -5.676 (17.9077)
  Week 24 (n=159, 164, 155) | -4.232 (14.6688) | -0.768 (19.6396) | -3.623 (20.1695)
  Week 28 (n=160, 161, 153) | -1.660 (16.9498) | 0.421 (22.1540) | -2.888 (17.1272)
  Week 32 (n=160, 163, 151) | -1.961 (17.8059) | 1.776 (21.1586) | -1.030 (19.2558)
  Week 36 (n=158, 160, 151) | -1.731 (16.7500) | 2.858 (20.9376) | 0.035 (20.9409)
  Week 40 (n=160, 160, 151) | -0.378 (17.4848) | 2.412 (20.8940) | -0.037 (20.6483)
  Week 44 (n=160, 158, 150) | 1.677 (17.2021) | 2.334 (21.0440) | 0.598 (19.6207)
  Week 48 (n=157, 157, 148) | -0.634 (16.2926) | 2.413 (22.0726) | -0.306 (19.0464)
  Week 52 (n=155, 154, 145) | -0.374 (17.5598) | 2.993 (20.3400) | -0.621 (16.9016)

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
percent change
  Week 4 (n=165, 170, 167) | -3.347 (9.1943) | -6.381 (9.8008) | -3.386 (9.8537)
  Week 8 (n=164, 168, 165) | -3.510 (9.3764) | -7.294 (9.7792) | -3.711 (11.0426)
  Week 12 (n=163, 168, 161) | -4.918 (9.1307) | -7.316 (9.7382) | -5.300 (10.5662)
  Week 16 (n=163, 167, 161) | -4.489 (10.9503) | -7.131 (10.7158) | -5.027 (12.2383)
  Week 20 (n=162, 166, 157) | -5.310 (10.0187) | -6.543 (10.2848) | -5.421 (11.6463)
  Week 24 (n=159, 164, 155) | -4.503 (9.5968) | -4.824 (11.2452) | -4.241 (13.3773)
  Week 28 (n=160, 161, 153) | -2.590 (11.5574) | -4.691 (11.0348) | -3.644 (11.0906)
  Week 32 (n=160, 163, 151) | -2.201 (11.0082) | -3.427 (11.2990) | -2.939 (11.0774)
  Week 36 (n=158, 160, 151) | -2.418 (10.7162) | -2.439 (11.0752) | -1.980 (12.9512)
  Week 40 (n=160, 160, 151) | -1.755 (10.7847) | -3.085 (10.7054) | -2.947 (12.9953)
  Week 44 (n=160, 158, 150) | -1.073 (10.0091) | -2.956 (9.9486) | -2.509 (12.1363)
  Week 48 (n=157, 157, 148) | -2.581 (9.8592) | -3.435 (11.1554) | -2.406 (11.8012)
  Week 52 (n=155, 154, 145) | -2.066 (10.9462) | -2.801 (11.0523) | -2.808 (10.6534)

9. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein - Cholesterol (HDL-C)
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
percent change
  Week 4 (n=165, 170, 167) | 0.849 (12.2814) | 2.184 (12.6361) | -0.762 (11.4762)
  Week 8 (n=164, 168, 165) | 1.886 (13.6679) | 1.298 (12.8820) | -0.955 (12.9760)
  Week 12 (n=163, 168, 161) | 0.535 (12.5694) | 1.085 (13.1746) | -0.561 (12.7619)
  Week 16 (n=163, 167, 161) | 1.276 (13.3975) | 1.699 (12.4080) | -0.134 (12.7453)
  Week 20 (n=162, 166, 157) | 2.708 (14.7306) | 2.913 (13.3232) | 1.034 (14.0619)
  Week 24 (n=159, 164, 155) | 4.569 (14.8251) | 5.684 (14.7141) | 2.693 (14.7185)
  Week 28 (n=160, 161, 153) | 4.712 (16.0076) | 6.117 (15.5220) | 2.975 (15.7048)
  Week 32 (n=160, 163, 151) | 6.456 (16.2378) | 6.890 (14.6459) | 3.012 (14.6151)
  Week 36 (n=158, 160, 151) | 8.234 (15.8749) | 8.516 (14.2641) | 4.946 (15.6107)
  Week 40 (n=160, 160, 151) | 8.410 (18.0364) | 8.359 (15.6201) | 5.264 (15.6110)
  Week 44 (n=160, 158, 150) | 7.983 (15.5313) | 7.182 (15.7227) | 4.533 (14.3921)
  Week 48 (n=157, 157, 148) | 6.191 (14.7070) | 7.144 (15.1433) | 4.499 (14.6233)
  Week 52 (n=155, 154, 145) | 6.738 (15.3629) | 6.932 (16.1796) | 5.183 (14.7508)

10. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein - Cholesterol
Description: Non-high-density lipoprotein cholesterol was calculated by subtracting high-density lipoprotein cholesterol from total cholesterol.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Number analyzed (Participants) | 165 | 171 | 167
percent change
  Week 4 (n=165, 170, 167) | -4.406 (11.2322) | -8.831 (12.2172) | -3.885 (12.3062)
  Week 8 (n=164, 168, 165) | -4.836 (11.6718) | -9.663 (11.6911) | -4.185 (13.9301)
  Week 12 (n=163, 168, 161) | -6.355 (11.1879) | -9.665 (11.8662) | -6.301 (12.7396)
  Week 16 (n=163, 167, 161) | -5.929 (13.2860) | -9.674 (13.2498) | -6.102 (15.3247)
  Week 20 (n=162, 166, 157) | -7.329 (12.1200) | -9.169 (12.6390) | -6.941 (14.3629)
  Week 24 (n=159, 164, 155) | -6.911 (11.1228) | -7.769 (13.3944) | -5.842 (15.4628)
  Week 28 (n=160, 161, 153) | -4.396 (13.6832) | -7.643 (13.3578) | -5.219 (13.4854)
  Week 32 (n=160, 163, 151) | -4.373 (13.3296) | -6.273 (14.3110) | -4.186 (13.7872)
  Week 36 (n=158, 160, 151) | -5.256 (13.2490) | -5.515 (14.4721) | -3.574 (16.2259)
  Week 40 (n=160, 160, 151) | -4.285 (14.7340) | -6.397 (14.1767) | -4.907 (16.5866)
  Week 44 (n=160, 158, 150) | -3.270 (12.4442) | -5.801 (13.3310) | -4.134 (15.6056)
  Week 48 (n=157, 157, 148) | -4.796 (12.2273) | -6.497 (14.6818) | -4.088 (15.0735)
  Week 52 (n= 155, 154, 145) | -4.340 (13.7408) | -5.255 (14.9219) | -4.830 (13.5956)

ADVERSE EVENTS:
Time Frame: Collection of AEs commenced from the time that the participant was first administered investigational product (Week 0) until the completion of study treatment (52 weeks of administration)
Description: At each study visit, the investigator or subinvestigator assessed whether any AEs had occurred. A neutral question, such as "How have you been feeling since your last visit?" asked. Participants reported AEs occurring at any other time during the study.
Arm/Group | TAK-085 2 g | TAK-085 4 g | EPA-E 1.8 g
Serious Adverse Events (participants affected / at risk) | 5/165 | 10/171 | 7/167
Other Adverse Events (participants affected / at risk) | 96/165 | 94/171 | 104/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 2 g (N=165) | TAK-085 4 g (N=171) | EPA-E 1.8 g (N=167)
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Neurogenic shock (Vascular disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-085 2 g (N=165) | TAK-085 4 g (N=171) | EPA-E 1.8 g (N=167)
Nasopharyngitis (Infections and infestations) | 57 | 43 | 42
Pharyngitis (Infections and infestations) | 14 | 15 | 15
Bronchitis (Infections and infestations) | 9 | 7 | 9
Seasonal allergy (Immune system disorders) | 6 | 6 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 9 | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 12 | 19 | 14
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 9
Dental caries (Gastrointestinal disorders) | 2 | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 12
Blood creatine phosphokinase increased (Investigations) | 13 | 7 | 18
Liver function test abnormal (Investigations) | 10 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.